CLINICAL TRIAL: NCT07136389
Title: An Open-label, Non-comparative Clinical Study of the Safety, Pharmacokinetics, Immunogenicity BCD-256 and Divozilimab in Monotherapy and Combination Therapy With Single and Multiple Intravenous Administration to Subjects With Systemic Lupus Erythematosus
Brief Title: Safety, Pharmacokinetics, Immunogenicity BCD-256-1 and Divozilimab in Subjects With Systemic Lupus Erythematosus
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BCD-256-1
Record Dates: First submitted 2025-08-08; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-06

CONDITIONS: Systemic Lupus Erthematosus
Keywords: divozilimab; anti-BDCA2; anti-CD20

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- BCD-256 Cohort 1 (Experimental)
  Interventions: Drug: BCD-256
- BCD-256 Cohort 2 (Experimental): Given satisfactory tolerability (no DLT events in all cohort 1 subjects for 14 days from the start of BCD-256 therapy), the subjects are included at the second dose level.
  Interventions: Drug: BCD-256
- BCD-256 Cohort 3 (Experimental): Given satisfactory tolerability (no DLT events in all cohort 2 subjects for 14 days from the start of therapy), the subjects are included at the third dose level.
  Interventions: Drug: BCD-256
- Divozilimab Cohort 4 (Experimental): The inclusion of subjects in Cohort 4 occurs in parallel with the enrollment of subjects in cohorts 1-3.
  Interventions: Drug: Divozilimab
- Divozilimab Cohort 5 (Experimental): The inclusion of subjects in Cohort 5 occurs in parallel with the enrollment of subjects in cohorts 1-3.
  Interventions: Drug: Divozilimab; Drug: BCD-256
- Cohort A (Experimental): Subjects will receive BCD-256 plus divozilimab
  Interventions: Drug: Divozilimab; Drug: BCD-256
- Cohort B (Experimental): Subjects will receive BCD-256 plus divozilimab
  Interventions: Drug: Divozilimab; Drug: BCD-256
- Cohort C (Experimental): Subjects will receive BCD-256 plus divozilimab
  Interventions: Drug: Divozilimab; Drug: BCD-256
- Cohort D (Experimental): Subjects will receive BCD-256 plus divozilimab
  Interventions: Drug: Divozilimab; Drug: BCD-256

INTERVENTIONS:
Drug: BCD-256 — Anti-BDCA2 human monoclonal antibody, concentrate for solution for infusion intravenously
  Other Names: Anti-BDCA2
  Arms: BCD-256 Cohort 1
Drug: BCD-256 — Anti-BDCA2 human monoclonal antibody, concentrate for solution for infusion intravenously
  Other Names: Anti-BDCA2
  Arms: BCD-256 Cohort 2
Drug: BCD-256 — Anti-BDCA2 human monoclonal antibody, concentrate for solution for infusion intravenously
  Other Names: Anti-BDCA2
  Arms: BCD-256 Cohort 3
Drug: Divozilimab — Ant-CD0 human monoclonal antibody, Concentrate for solution for infusion intravenously
  Other Names: Anti-CD20
  Arms: Cohort A; Cohort B; Cohort C; Cohort D; Divozilimab Cohort 4; Divozilimab Cohort 5
Drug: BCD-256 — Anti-BDCA2 human monoclonal antibody, concentrate for solution for infusion intravenously
  Other Names: Anti-BDCA2
  Arms: Cohort A; Cohort B; Cohort C; Cohort D; Divozilimab Cohort 5

SUMMARY:
The goal of this clinical trial to investigate the safety, pharmacokinetics, pharmacodynamics, immunogenicity, and preliminary efficacy of BCD-256 alone and in combination with anti-CD20 therapy (divozilimab) as second- or later-line therapy in subjects with skin lesions due to mild to moderate systemic lupus erythematosus. The study consists of the first stage (cohorts 1-5) and the second stage (cohorts A - D).

DETAILED DESCRIPTION:
The study is conducted in 2 stages which involve different subjects. Stage 1 of the study have a modified "3+3" design and involves dose escalation of BCD-256 in 1-3 cohorts with an interval of at least 14 days dose - limiting toxicicity (DLT) (DLT assessment period) between cohorts 1-3. In cohorts 4 and 5, the administration of divozilimab is carried out in parallel with cohorts 1-3. A decision on the possibility of starting Stage 2 and including new subjects in it will be made after approval by thethe Cohort Dosing Safety Committee (CDSC) of an interim report (for 12 weeks of therapy). Stage 2 of the study will involve the use of BCD-256 in combination with divozilimab in 4 cohorts, BCD-256 dose levels in cohorts will be determined based on the results of the main period of Stage 1 (for 12 weeks of therapy).

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent to participate in the study and the subject's ability to comply with the requirements of the clinical study protocol.
2. Age from 18 to 70 years at the time of signing the informed consent form.
3. Body weight from 45 kg, BMI of 18 to 30 kg/m2.
4. Diagnosed with SLE in accordance with at least 4 classification criteria of SLICC (2012), including 1 clinical sign or 1 immunological manifestation.
5. Disease activity according to the SLEDAI score of 6-12.
6. CLASI-A ≥ 9 at screening, at least one skin lesion with R-CLASI ≥ 6 at screening.
7. Positive test for antinuclear antibodies at screening (titer ≥ 1:160) and/or increased level of double-stranded DNA antibody (≥ 2 ULN).
8. History of the disease ≥24 weeks at the time of signing the informed consent form.
9. Active skin disease according to the CLASI scale, despite the use of topical and systemic glucocorticoids and/or antimalarial drugs for at least 3 months at the time of signing the informed consent form.
10. Women of childbearing potential have a negative pregnancy test at screening.
11. Willingness of men and women of childbearing potential to use two highly effective contraception methods from the signing of the informed consent form, throughout the study and for 6 months after the administration of the last product dose. In this study, a woman is considered to be of childbearing potential if she is postmenarcheal, did not reach menopause (amenorrhea for ≥12 months, which cannot be explained by any other cause than menopause), and did not undergo surgical sterilization (removal of ovaries, fallopian tubes, and/or uterus).

Exclusion Criteria:

1. Presence of active lupus nephritis or chronic kidney disease (urine protein to creatinine ratio >2.0 or estimated glomerular filtration rate < 30 mL/min/1.73m2).
2. A history of CNS associated with SLE, involvement including, but not limited to, the following symptoms: seizures, impaired consciousness, psychosis, delirium or confusion, aseptic meningitis, ascending or transverse myelitis, chorea, cerebellar ataxia, multiple mononeuritis, or demyelinating syndromes.
3. The presence of uncontrolled neuropsychiatric disorders, severe depression and/or suicide attempts at the time of signing the ICF or within 1 year prior to signing the informed consent form, as well as the risk of suicide and/or any mental illness as assessed by the investigator.
4. A history of antiphospholipid syndrome.
5. Use of the following groups of drugs before signing ICF:

   * abatacept, belimumab, tocilizumab or tumor necrosis factor (TNF) inhibitors within 3 months or 5 half-lives prior to screening (whichever is longer);
   * rituximab, atacicept, ocrelizumab or other biological agents targeting B cells within 9 months prior to screening;
   * cyclosporine, tacrolimus, pimecrolimus, sirolimus, imiquimod, intravenous immunoglobulin, intravenous and oral cyclophosphamide, and plasmapheresis within 3 months prior to screening;
   * thalidomide or lenalidomide within 2 months prior to screening;
   * receiving oral glucocorticoids at a dose of > 20 mg /day in terms of prednisone or dose changes for at least 4 weeks prior to screening;
   * other immunosuppressive or disease modifying treatments for SLE under at least one of the following conditions:

     1. the drugs were started less than 3 months before screening,
     2. the dose was changed within 1 month prior to screening,
     3. the medications were taken in doses exceeding the specified amounts: antimalarial drugs (hydroxychloroquine up to 6.5 mg/kg/day, quinacrine up to 5 mg/kg/day, chloroquine 3 mg/kg/day), dapsone 150 mg/day, methotrexate 20 mg/week, azathioprine 200 mg/day, 6-mercaptopurine 1.5 mg/kg/day, and mycophenolate mofetil 2 g/day or mycophenolate sodium 1440 mg/day.
6. Laboratory test values:

   * absolute neutrophil count <1,500/µL (1.5×109/L);
   * lymphocyte count <800/µL cells×109/L (0.8×109/L);
   * platelets <75,000/µL (75×109/L);
   * hemoglobin ≤ 9 g/dL (≤ 90 g/L);
   * serum creatinine >1.5×ULN, OR for subjects with a creatinine level >1.5×ULN, creatinine clearance/glomerular filtration rate <30 mL/min ;
   * total bilirubin > 1.5 × ULN (for subjects with Gilbert's syndrome, total bilirubin levels should not exceed 50 µmol/L);
   * AST or ALT >2×ULN;
   * alkaline phosphatase >2×ULN.
7. Concomitant diseases and/or conditions that significantly increase the risk of AEs during the study:

   * uncontrolled hypertension (subjects with arterial hypertension not controlled by 3 antihypertensive drugs (SBP ≥ 140 mmHg or DBP ≥ 90 mmHg));
   * stable angina pectoris, functional class III-IV according to the Canadian Cardiovascular Society, CCS;
   * acute coronary syndrome less than 6 months before the start of therapy in the study;
   * congestive heart failure (NYHA III-IV);
   * clinically significant arrhythmia at the opinion of the investigator that are not amenable to the maximum possible antiarrhythmic therapy (therapy should be stable for 4 weeks before the first dose of BCD 256/divozilimab);
   * moderate or severe asthma, stage III-IV chronic obstructive pulmonary disease, history of angioneurotic edema, severe respiratory failure;
   * any other concomitant disease or condition, which, in the Investigator's opinion, significantly increases the risk of AEs in the study.
8. Any active skin diseases other than SLE that may interfere with the study and effect assessment (e.g., psoriasis, drug-induced lupus, vitiligo, rosacea, local skin infections).
9. Documented presence of one or more systemic concomitant diseases requiring systemic glucocorticoid therapy (e.g., asthma, IBD, psoriasis, acute uveitis). Oral, rectal or any injectable route of administration will be considered systemic.

   Exception: concomitant diseases requiring the use of glucocorticoids by other methods of administration (for example, topical, inhalation, intranasal, into the conjunctival sac, etc.) are allowed. Subjects with endocrinopathy requiring only hormone replacement therapy are also eligible.
10. A history of herpes infection: herpes encephalitis, ocular herpes, and disseminated herpes infection.
11. Documented diagnosis of chickenpox, cytomegalovirus infection, infectious mononucleosis, herpes zoster, genital herpes, herpetic gingivostomatitis within 3 months before signing the ICF and during the screening period.
12. A current diagnosis or a history of a severe immunodeficiency of any origin.
13. A history of or active or latent tuberculosis (positive Diaskintest®, QuantiFERON or T-SPOT.TB test, in the absence of signs of pulmonary tuberculosis on chest X-ray or CT). Subjects who have ongoing social contacts with active tuberculosis should also not be included in the clinical study.
14. A documented diagnosis of any other chronic infection that, in the opinion of the investigator, can increase the risk of infectious complications .
15. Active infectious diseases (requiring hospitalization, parenteral use of antibacterial, antimycotic or antiprotozoal drugs) within 8 weeks prior to signing the ICF and during the screening period.
16. Systemic antibacterial, antimycotic or antiprotozoal therapy within 8 weeks prior to signing the ICF and during the screening period.
17. Scheduled vaccination with live, live attenuated vaccines or non-live vaccines within 1 month prior to screening and throughout the study, and within 4 months after the last dose of the study drug or divozilimab.
18. Established HIV infection, hepatitis B, active hepatitis C .
19. COVID-19, major surgery within 4 weeks prior to signing the ICF or major surgery planned for the period of participation in the study.
20. Simultaneous participation in other clinical studies, as well as previous participation in other clinical studies less than 3 months before signing the ICF, prior participation in the main period of this study.

    Exception: subjects who dropped out of this study at screening.
21. Comorbidities (including, but not limited to, metabolic, hematological, renal, hepatic, pulmonary, neurological, endocrine, cardiac, infectious, gastrointestinal disorders), including disorders ongoing at the time of screening, which, in the opinion of the investigator, may affect the course of SLE, the results of assessment of its symptoms, or create an unacceptable risk to the subject from study therapy.
22. Lymphoproliferative diseases or solid tumors (including basal cell carcinoma in situ) with a remission duration of less than 5 years, except for cured cervical cancer in situ.
23. Impossibility of intravenous administration of drugs.
24. Hypersensitivity or allergy to any of the components of BCD-256 and divozilimab. A history of severe allergic, anaphylactic or other hypersensitivity reactions to chimeric or humanized antibodies or hybrid proteins.
25. Pregnancy or breastfeeding, or planning pregnancy or fatherhood throughout the study and for 6 months after the last dose of the drug.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with adverse events | 85 days
Proportion of subjects with serious adverse events | 85 days
Proportion of subjects with treatment-related adverse events | 85 days
Proportion of subjects with CTCAE 5.0 grade ≥ 3 adverse events | 85 days
Proportion of cases of early discontinuation of study therapy due to adverse events | 85 days
Proportion of subjects with adverse events of special interest | 85 days

SECONDARY OUTCOMES:
Time to Reach Maximum Observed Concentration (Tmax) in the first cycle of therapy | 0-15 days
Terminal Elimination Half-Life (t1/2) in the first cycle of therapy | 0-15 days

OTHER OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 to ending at the last measured concentration at time t (AUC0-t) in the first cycle of therapy | 0 -15 days
Area Under the Concentration-Time Curve from Time 0 Extrapolated to Infinity (AUC0-∞) in the first cycle of therapy | 0 - 15 days
Area Under the plasma-concentration versus time curve (AUC) over one dosing interval (τ) when steady-state (ss) conditions have been reached, representing the average drug exposure during that interval n the third cycle of therapy | 57 - 85 days
Maximum Observed Concentration (Cmax) in the first cycle of therapy | 0 -15 days
Trough concentation (Ctroug) in the first and second cycle of therapy | 0 - 57 days

CONTACTS AND LOCATIONS:
Overall Officials: Arina V Zinkina-Orikhan, PhD, Study Director — Director of Clinical Development Department, BIOCAD
Locations (1):
- "Multidisciplinary medical center for adults and children №157", Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials | BIOCAD — https://ct.biocad.ru/en/nozology?utm_source=biocad.ru&utm_medium=referral&utm_campaign=biocad_referral&utm_reffere=biocad.ru